CLINICAL TRIAL: NCT05715749
Title: Exploring the Feasibility and Utility of In-home Body Weight Support Harness System Use in Children Treated for Spinal Muscular Atrophy: a Pilot Study
Brief Title: Body Weight Support Harness System in Spinal Muscular Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Megan Iammarino, Research Physical Therapist, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB18-00484
Record Dates: First submitted 2023-01-20; First posted 2023-02-08 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Spinal Muscular Atrophy Type I; Spinal Muscular Atrophy Type II
Keywords: exercise; physical therapy
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood; Motor Activity | interventions — bbc3 protein, zebrafish

STUDY DESIGN:
Masking Description: Outcomes assessors are masked to previous participant performance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- In-home body weight support harness system (Experimental): All participants will be entered into treatment arm and receive an in-home body weight support harness system
  Interventions: Other: In-home body weight support harness system

INTERVENTIONS:
Other: In-home body weight support harness system — A portable, adjustable body weight support harness system that occupies roughly 9 feet x 9 feet space in the home. The system allows 360 degrees of mobility anywhere within the footprint of the frame. The amount of body weight support is adjustable.
  Other Names: The Portable Mobility Aid for Children (PUMA)

SUMMARY:
The goal of this pilot interventional study is to learn about the use of an in-home harness system in children who have been treated for spinal muscular atrophy. The main questions it aims to answer are:

1. Is the in-home body weight support harness system a feasible option for families to use?
2. Is the in-home body weight support harness system a useful tool for children treated for spinal muscular atrophy?
3. Is the in-home body weight support harness system a safe tool for children treated for spinal muscular atrophy?

Participants will be given an in-home body weight support harness system and taught how to use it. Families will document how often and for how long they use the system over 6 months. Children will be given tests of motor function at the beginning, 3-months, and 6-months. At the end of the study, families will be asked to fill out a questionnaire about thier experience using the system.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed heterozygous mutation in SMN1 gene and 2 or 3 copies of SMN2 (historically, SMA Type 1 and Type 2)
* Past or current treatment with nusinersen, onasemnogene abeparvovec, or risdiplam
* Upright head control (defined as the ability to lift head from full forward flexion)
* Weight under or 50lbs
* Confirmed motor delay

Exclusion Criteria:

* 4+ copies of SMN2 (historically, SMA Type 3 and 4)
* Evidence of lower limb injury or recent fracture
* In the opinion of the investigator, it was unsafe for the child to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Caregiver survey | End of study visit (month 6)
  A five question likert-style survey asking families to rate their experience during the study. The scales asks the family to rate (1) the perceived impact of BWSS on motor and (2) non-motor skills, (3) the child's perceived enjoyment using the system, (4) the ease of equipment use, and (5) if the family believed that use of the BWSS was beneficial on a 5-point Likert scale; scores of 4 or 5 were considered favorable, scores of 3 were considered neutral, and scores of 1 or 2 were considered unfavorable. Higher scores indicate greater perceived benefit of participation.
Change in The Neuromuscular Gross Motor Outcome (GRO) scale | Completed at baseline, 3 months, and 6 months
  A 50-item performance-based outcome developed to quantify motor function across the span of age and abilities in individuals with neuromuscular disorders including spinal muscular atrophy (SMA). Scores range from 0 - 100 points; higher scores reflect a greater level of function. An increase in score indicates a better outcome.
Change in Hammersmith Functional Motor Scale Expanded (HFMSE) | Completed at baseline, 3 months, and 6 months
  A disease-specific and performance-based outcomes originally developed to measure motor skill in untreated individuals with SMA. Scores range from 0 - 66 points; higher scores reflect a greater level of function. An increase in score indicates a better outcome.
Change in Revised Hammersmith Scale (RHS) | Completed at baseline, 3 months, and 6 months
  A disease-specific and performance-based outcomes originally developed to measure motor skill in untreated individuals with SMA, revised following Rasch analysis of HFMSE. Scores range from 0 - 69 points; higher scores reflect a greater level of function. An increase in score indicates a better outcome.
Change in Bayley Scales of Infant and Toddler Development 3rd ed. (Bayley-III), Gross motor subtest | Completed at baseline, 3 months, and 6 months
  A norm-referenced developmental assessment of gross motor skill in children 16 days - 3.5 years of age. Raw scores range from 0 - 72. Higher scores indicate a greater level of funcion. An increase in score indicates a better outcome.
Change in World Health Organization Motor Milestone Checklist | Completed at baseline, 3 months, and 6 months
  A checklist of key gross motor milestones expected during typical development. Scores can range from 0 - 6 milestones achieved. Achievement of a greater number of milestones indicates better outcomes.

SECONDARY OUTCOMES:
Harness use log | Completed throughout 6-month study period
  A log to document frequency (each use) and duration (how long it was used at one time) of harness system use.

CONTACTS AND LOCATIONS:
Overall Officials: Megan A Iammarino, DPT, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will be provided in summary form at manuscript submission. Certain individual participant data will be available in manuscript as well.

REFERENCES:
- [Derived] Iammarino MA, Alfano LN, Reash NF, Sabo B, Conroy S, Noritz G, Wendland M, Lowes LP. Feasibility and utility of in-home body weight support harness system use in young children treated for spinal muscular atrophy: A single-arm prospective cohort study. PLoS One. 2024 Mar 19;19(3):e0300244. doi: 10.1371/journal.pone.0300244. eCollection 2024. PMID 38502672